CLINICAL TRIAL: NCT07370493
Title: A Multicenter, Retrospective Analysis to Evaluate Radiographic Outcomes and Safety Profiles Along Prospective Follow-Up Periods for Patients Implanted With 2 Levels of Prodisc® C Vivo Devices.
Brief Title: Retrospective Analysis of Patients Implanted With 2 Levels of Prodisc® C Vivo Devices
Status: Enrolling by invitation | Type: Observational
Sponsor: Centinel Spine (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Other Study IDs: VAL-P-0190
Record Dates: First submitted 2025-11-13; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Degenerative Disc Disease; Cervical Spine Degenerative Disease; Symptomatic Cervical Disc Disease; Cervical Spine Degenerative Disc Disease
Keywords: Degenerative disc disease; cervical spine degenerative disc disease; Cervical Total Disc Arthroplasty; Symptomatic Cervical Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Retrospective chart review: Retrospective chart review of patients treated with prodisc® C Vivo at 2 contiguous levels.
  Interventions: Device: Prodisc C Vivo
- Prospective follow-up: Prospective follow-up of patients treated with prodisc® C Vivo at 2 contiguous levels.
  Interventions: Device: Prodisc C Vivo

INTERVENTIONS:
Device: Prodisc C Vivo — The prodisc® C Vivo device is a non-keeled cervical disc replacement prosthesis. The device is modular intervertebral disc prostheses designed to replace a diseased and/or a degenerated disc of the cervical spine in SCDD patients, thereby restoring disc height, biomechanical stability and allowing the potential for motion at the affected vertebral segment.

SUMMARY:
The objective of the study is to evaluate the safety and post-operative performance profile of the prodisc® C Vivo after implantation in comparison to the relevant clinical literature.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate (estimate) the post-operative performance of prodisc® C Vivo overall, after implantation. Post-operative device performance will be estimated using Patient Reported Outcomes (PROs) and radiographic data derived from the patient's surgical charts and medical history.

The secondary objectives of this study are to assess:

* patients with no secondary surgical interventions (SSIs), i.e. revision, removal, re-operation, supplemental fixation at the index level(s)
* the rates of ADEs inclusive of intraoperative and post-operative complications
* Patient Reported Outcomes (PROs)
* Outcome self-assessment of Health Survey (SF 12 or 36 as available)

ELIGIBILITY:
Inclusion Criteria:

* In order for a patient's data to be included in this study, he/she has to meet the indications and not possess any of the specific or general contraindications listed in the Instructions For Use (IFU).
* They must provide written informed consent with appropriate documentation noted in source documentation (prospective cohort only).

Exclusion Criteria:

-There are no additional exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients treated with prodisc® C Vivo implants at 2 levels in the cervical spine for the treatment of SCDD.
  Patients who underwent the initial surgery with the device, from 2010 until 2024 will be considered eligible for this study.
  Patients who are excluded from this study and their reason will be noted.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the Occurrence of Secondary Surgical Interventions in Patients Treated with prodisc® C Vivo at 2 Levels | 10 year post-operative screening of prodisc C Vivo patients implanted from JAN 2010 to present
  The primary objective of the study is to evaluate the post-operative performance of the prodisc® C Vivo after implantation by the occurrence of secondary surgical interventions in patients treated with prodisc® C Vivo at 2 levels. The State of the Art (SOTA) will be used as the comparison data collected in this study.

SECONDARY OUTCOMES:
Assessment to demonstrate the continuous clinical and radiographic status of the prodisc C Vivo implants allowing characterization of performance of the device by nominal variables (percentages) based on ADEs, SSIs, PROs, and SF 12 data collection | 10 Year Post-operative 10 year post-operative screening of prodisc C Vivo patients implanted from JAN 2010 to present
  Nominal variables will be presented as count (percent). For numerical variables, the results will be presented as minimum, 25th percentile, mean, standard deviation, median, 75th percentile and maximum. Frequency tables for system organ class and preferred terms will be compiled based on participants experiencing an ADE (Adverse Device Event), and on the number of ADEs (from initial surgery to present, including intraoperative and post-operative complications). These percentage variables will include multiple data collection factors, such as the number and proportions of patients with no secondary surgical interventions (SSIs) (revision, removal, re-operation, supplemental fixation) at the index level(s) from initial surgery to present, Patient Reported Outcome (PRO) assessments, and self-assessment of Health Surveys (SF 12).

CONTACTS AND LOCATIONS:
Overall Officials: James Kuras, MS, Study Director — Centinel Spine
Locations (1):
- ONZ Spine, Recklinghausen, Germany

IPD SHARING:
Plan to Share IPD: No